CLINICAL TRIAL: NCT05067335
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of Romosozumab Treatment in Postmenopausal Chinese Women With Osteoporosis
Brief Title: A Study to Test the Efficacy, Safety and Tolerability of Romosozumab Treatment in Postmenopausal Chinese Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OP0002
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Phase 3; Chinese Patients; Romosozumab
MeSH Terms: conditions — Osteoporosis | interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Romosozumab (Experimental): Subjects randomized to this arm will receive romosozumab during all treatment Periods.
  Interventions: Drug: Romosozumab
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo during the Double-Blind-Placebo controlled Period and romosozumab during the Open-Label treatment Period
  Interventions: Drug: Romosozumab; Drug: Placebo

INTERVENTIONS:
Drug: Romosozumab — Subjects will receive romosozumab in a specified sequence during the treatment Period.
Drug: Placebo — Subjects will receive Placebo in a specified sequence during the treatment Period.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect of treatment with romosozumab for 6 months compared with placebo on the percent changes in bone mineral density (BMD) at the lumbar spine, at the total hip and femoral neck in postmenopausal Chinese women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is considered reliable and capable of adhering to the protocol, visit schedule, and medication intake according to the judgment of the investigator
* Subject is an ambulatory postmenopausal Chinese women, 55 to 90 years of age (inclusive) at the time of Screening. Postmenopause is defined as no spontaneous vaginal bleeding or spotting for 12 or more consecutive months prior to Screening
* Subject has a bone mineral density (BMD) T-score ≤-2.50 at the lumbar spine, total hip, or femoral neck, as assessed by the central imaging vendor at the time of Screening based on DXA scans, and using data for Caucasian women from the National Health and Nutritional Examination Survey (NHANES, 1998)
* Subject must have at least 1 of following independent risk factors for fracture:

  * History of fragility fracture (except hip fracture, a severe vertebral fracture or more than 2 moderate vertebral fractures)
  * Parental history of hip fracture
  * Low body weight (body mass index ≤19kg/m2)
  * Elderly (age ≥ 65 years)
  * Current smoker
* Subject has at least 2 vertebrae in the L1 to L4 region and at least 1 hip that are evaluable by dual-energy x-ray absorptiometry (DXA), as assessed by the central imaging vendor

Exclusion Criteria:

* Subject has a BMD T-score of ≤-3.50 at the total hip or femoral neck, as assessed by the central imaging vendor at the time of Screening based on DXA scans, and using data for Caucasian women from NHANES 1998
* Subject has a known history of hip fracture
* Subject has any severe (SQ3) or more than 2 moderate (SQ2) vertebral fractures, as assessed by the central imaging vendor based on the lateral spine x-ray at Screening
* Subject has a history of myocardial infarction (MI)
* Subject has a history of stroke
* Subject has a vitamin D insufficiency, defined as 25 (OH) vitamin D levels <20 ng/mL, as assessed by the central laboratory at Screening. Vitamin D repletion will be permitted and the subject may be retested once within the Screening Period
* Subject has used oral bisphosphonates:

  * Any doses received within 3 months prior to randomization
  * More than 1 month of cumulative use between 3 and 12 months prior to randomization
  * More than 3 years of cumulative use, unless the last dose was received ≥5 years prior to randomization
* Subject has used intravenous (iv) bisphosphonates:

  * zoledronic acid

    * Any doses received within 3 years prior to randomization
    * More than 1 dose received within 5 years prior to randomization
  * iv ibandronate, iv pamidronate, or iv alendronate (ALN)

    * Any doses received within 12 months prior to randomization
    * More than 3 years of cumulative use, unless the last dose was received ≥5 years prior to randomization
* Subject has used denosumab or any cathepsin K inhibitor:

  ● Any doses received within 18 months prior to randomization
* Subject has used tibolone, cinacalcet, or calcitonin:

  * Any doses received within 3 months prior to randomization
* Subject has used teriparatide (TPTD) or any parathyroid hormone (PTH) derivative:

  * Any doses received within 3 months prior to randomization
  * More than 1 month of cumulative use between 3 and 12 months prior to randomization
* Subject has used systemic oral or transdermal estrogen or selective estrogen receptor modulators (SERMs):

  ● More than 1 month of cumulative use within 6 months prior to randomization
* Subject has used strontium ranelate or fluoride:

  ● More than 1 month of cumulative use within 5 years prior to randomization
* Subject has used hormonal ablation therapy:

  ● More than 1 month of cumulative use within 6 months prior to randomization
* Subject has used systemic glucocorticosteroids:

  ● ≥5mg prednisone equivalent per day for more than 14 days within 3 months prior to randomization
* Subject has a history of osteonecrosis of the jaw (ONJ) or atypical femoral fracture (AFF)
* Subject has evidence of any of the following:

  1. Current, uncontrolled hyper- or hypothyroidism. Uncontrolled hyperthyroidism is defined as thyroid-stimulating hormone (TSH) and thyroxine (T4) outside of the normal range. Uncontrolled hypothyroidism is defined as TSH >10
  2. Current, uncontrolled hyperparathyroidism or history of hypoparathyroidism. Uncontrolled hyperparathyroidism is defined as PTH outside the normal range in subjects with concurrent hypercalcemia or PTH values >20 % above upper limit of normal (ULN) in normocalcemic subjects
  3. Current hypercalcemia or hypocalcemia, defined as albumin-adjusted serum calcium outside the normal range, as assessed by the central laboratory at the time of Screening. Albumin-adjusted serum calcium levels may be retested once in case of an elevated albumin-adjusted serum calcium level within 1.1xULN of the laboratory's reference ranges
  4. Subject has ≥3xULN of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (≥1.5xULN total bilirubin if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35 %)

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 327 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (30):
- China (30):
  - Op0002 20040, Beijing
  - Op0002 20115, Beijing
  - Op0002 20125, Beijing
  - Op0002 20127, Beijing
  - Op0002 20128, Beijing
  - Op0002 20130, Beijing
  - Op0002 20131, Beijing
  - Op0002 20157, Beijing
  - Op0002 20021, Chengdu
  - Op0002 20133, Chengdu
  - Op0002 20137, Chengdu
  - Op0002 20205, Foshan
  - Op0002 20117, Guangzhou
  - Op0002 20124, Guangzhou
  - Op0002 20209, Nanchang
  - Op0002 20135, Nanjing
  - Op0002 20202, Pingxiang
  - Op0002 20199, Rui’an
  - Op0002 20116, Shanghai
  - Op0002 20118, Shanghai
  - Op0002 20121, Shanghai
  - Op0002 20123, Shanghai
  - Op0002 20129, Shanghai
  - Op0002 20119, Suzhou
  - Op0002 20204, Suzhou
  - Op0002 20122, Tianjin
  - Op0002 20136, Tianjin
  - Op0002 20120, Wuhan
  - Op0002 20134, Yueyang
  - Op0002 20132, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in October 2021 and concluded in November 2023.
Pre-assignment Details: Participant flow refers to the Randomized Set.
Groups:
- Placebo: Participants randomized to this arm received a matching placebo subcutaneously (sc) every month (QM) during the 6-month Double-blind (DB) Period.
- Romosozumab: Participants randomized to this arm received romosozumab (Romo) 210 milligrams (mg) sc QM during the 6-month Double-blind Period.
- Placebo/Romosozumab: After completion of the 6-month Double-blind Period, participants initially randomized to placebo arm switched to receive romosozumab 210 mg sc QM during the 6-month Open-label (OL) Period (up to Month 12).
- Romosozumab/Romosozumab: After completion of the 6-month Double-blind Period, participants initially randomized to romosozumab arm continued to receive romosozumab 210 mg sc QM during the Open-label Period (up to Month 12).
Period: Double-blind Period: Day 1 - Month 6
Arm/Group | Placebo | Romosozumab | Placebo/Romosozumab | Romosozumab/Romosozumab
Started | 109 | 218 | 0 | 0
Completed | 100 | 204 | 0 | 0
Not Completed | 9 | 14 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 10 | 0 | 0
Not completed — Patient Voluntary Withdrawal | 1 | 0 | 0 | 0
Not completed — The Patient Withdrew Early Due To Their Own Reasons | 0 | 1 | 0 | 0
Period: Open-label Period: Month 7 - 12
Arm/Group | Placebo | Romosozumab | Placebo/Romosozumab | Romosozumab/Romosozumab
Started | 0 | 0 | 99 (1 participant completed the Double-blind Period but withdrew due to an adverse event before starting the Open-label Period.) | 204
Completed | 0 | 0 | 93 | 199
Not Completed | 0 | 0 | 6 | 5
Not completed — Adverse Event | 0 | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — Subject Was Unable To Comply With Study Procedures Due To Prolonged Withdrawal From Medication | 0 | 0 | 1 | 0
Not completed — Did not receive Open-label IMP at Month 6 and then discontinued | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the RS which consisted of study participants who were randomized into this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romosozumab | Total
Number analyzed (Participants) | 109 | 218 | 327
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (6.1) | 67.0 (5.7) | 67.1 (5.8)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 yrs | 31 | 63 | 94
  65 - <85 yrs | 76 | 154 | 230
  >=85 yrs | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 218 | 327
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 109 | 218 | 327
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 109 | 218 | 327

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) at the Lumbar Spine to the End of Double-Blind Period
Description: Percent change from baseline in BMD at the lumbar spine was assessed by dual-energy x-ray absorptiometry (DXA) at 6 months. Missing postbaseline BMD other than due to COVID-19 were imputed using the last observation carried forward (LOCF) approach. Missing or out of window (exceed 70 days since previous IMP) post-baseline DXA BMD due to COVID-19 were set to missing and imputed by multiple imputation under missing at random approach. LSM = least square mean.
Time Frame: From Baseline (Day 1) to the end of the Double-blind Period (Month 6)
Population: The Full Analysis Set (FAS) consisted of all randomized study participants who received at least 1 dose of investigational medicinal product (IMP) and provided at least 1 Baseline and post-Baseline BMD measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 104 | 214
percent change | 0.44 (0.442) | 9.81 (0.323)
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; The ANCOVA model was used and included treatment group, Baseline DXA BMD value, machine type (hologic or lunar) at Baseline, age strata group (stratification factor), region, and interaction of Baseline DXA BMD value and machine type at Baseline as independent variables; Test type: Superiority; p < 0.001, ANCOVA; Difference in LSM(Romosozumab - Placebo) = 9.37, 95% CI 2-sided [8.34 to 10.39], Standard Error of Mean 0.524

2. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the Double-Blind Period
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a IMP, whether or not related to the IMP. TEAEs are defined as all AEs started on or worsened in severity on or after the date of receiving first dose of IMP and before or on the end of study (EOS) date.
Time Frame: From Baseline to the end of the Double-blind Period (Month 6)
Population: The Safety Set (SS) consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 109 | 218
percentage of participants | 70.6 | 72.9

3. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events for Romosozumab During Overall Period
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with use of a IMP, whether or not related to IMP. TEAEs are defined as all AEs started on or worsened in severity on or after date of receiving first dose of IMP and before or on EOS date except lipid-type AEs starting on date of first dose of IMP and not worsening (and not deemed IMP related by the investigator). As pre-specified in Protocol and SAP, TEAEs were assessed and reported for 6 months for participants in placebo/romosozumab arm (Open-label Period) and for a total of 12 months for participants in romosozumab/romosozumab arm (Double-blind Period + Open-label Period combined) + 3 months of Safety follow-up for both arms (Up to Month 15) during overall period.
Time Frame: From Month 7 up to Month 12 (Placebo/Romo) and From Day 1 up to Month 12 (Romo/Romo) + 3-month SFU (up to Month 15)
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP. The SS for open label period consisted of all randomized study participants who received at least 1 dose of IMP during open label period.
Measure: Number; unit: percentage of participants
Groups:
- Romosozumab/Romosozumab Overall: Participants who received romosozumab 210 mg sc QM during the 6-month Double-blind Period and continued to receive romosozumab 210 mg sc QM during the 6-month Open-label Period.
Arm/Group | Placebo/Romosozumab | Romosozumab/Romosozumab Overall
Number analyzed (Participants) | 98 | 218
percentage of participants | 80.6 | 88.1

4. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Total Hip to the End of Double-Blind Period
Description: Percent change from baseline in BMD at the total hip was assessed by DXA at 6 months. Missing postbaseline BMD other than due to COVID-19 were imputed using the LOCF approach. Missing or out of window (exceed 70 days since previous IMP) post-baseline DXA BMD due to COVID-19 were set to missing and imputed by multiple imputation under missing at random approach.
Time Frame: From Baseline to the end of the Double-blind Period (Month 6)
Population: The FAS consisted of all randomized study participants who received at least 1 dose of IMP and provided at least 1 Baseline and post-Baseline BMD measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 104 | 214
percent change | 0.07 (0.285) | 2.93 (0.206)
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Difference in LSM(Romosozumab - Placebo) = 2.86, 95% CI 2-sided [2.18 to 3.54], Standard Error of Mean 0.348

5. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Femoral Neck to the End of the Double-Blind Period
Description: Percent change from baseline in BMD at the femoral neck was assessed by DXA at 6 months. Missing postbaseline BMD other than due to COVID-19 were imputed using the LOCF approach. Missing or out of window (exceed 70 days since previous IMP) post-baseline DXA BMD due to COVID-19 were set to missing and imputed by multiple imputation under missing at random approach.
Time Frame: From Baseline to the end of the Double-blind Period (Month 6)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 104 | 214
percent change | -0.15 (0.406) | 3.33 (0.347)
Statistical Analysis 1: Comparison: Placebo vs Romosozumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Difference in LSM(Romosozumab - Placebo) = 3.48, 95% CI 2-sided [2.58 to 4.38], Standard Error of Mean 0.458

6. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Lumbar Spine at Month 12
Description: Percent change from Baseline in BMD at the lumbar spine was assessed by DXA at 12 months. Missing postbaseline BMD other than due to COVID-19 were imputed using the LOCF approach. Missing or out of window (exceed 70 days since previous IMP) post-baseline DXA BMD due to COVID-19 were set to missing and imputed by multiple imputation under missing at random approach. For Placebo/Romosozumab Treatment group, only the post Month 6 value was used for imputation for Open-label Period, the values in the Double-blind Period were not carried forward into the Open-label Period.
Time Frame: Baseline, Month 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo/Romosozumab Overall: Participants who received placebo during the 6-month Double-blind Period and switched to receive romosozumab 210 mg sc QM during the 6-month Open-label Period.
Arm/Group | Placebo/Romosozumab Overall | Romosozumab/Romosozumab Overall
Number analyzed (Participants) | 104 | 214
percent change | 8.80 (0.554) | 13.04 (0.389)

7. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Total Hip at Month 12
Description: Percent change from Baseline in BMD at the total hip was assessed by DXA at 12 months. Missing postbaseline BMD other than due to COVID-19 were imputed using the LOCF approach. Missing or out of window (exceed 70 days since previous IMP) post-baseline DXA BMD due to COVID-19 were set to missing and imputed by multiple imputation under missing at random approach. For Placebo/Romosozumab Treatment group, only the post Month 6 value was used for imputation for Open-label Period, the values in the Double-blind Period were not carried forward into the Open-label Period.
Time Frame: Baseline, Month 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo/Romosozumab Overall | Romosozumab/Romosozumab Overall
Number analyzed (Participants) | 104 | 214
percent change | 1.83 (0.306) | 4.22 (0.216)

8. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Femoral Neck at Month 12
Description: Percent change from Baseline in BMD at the femoral neck was assessed by DXA at 12 months. Missing postbaseline BMD other than due to COVID-19 were imputed using the LOCF approach. Missing or out of window (exceed 70 days since previous IMP) post-baseline DXA BMD due to COVID-19 were set to missing and imputed by multiple imputation under missing at random approach. For Placebo/Romosozumab Treatment group, only the post Month 6 value was used for imputation for Open-label Period, the values in the Double-blind Period were not carried forward into the Open-label Period.
Time Frame: Baseline, Month 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo/Romosozumab Overall | Romosozumab/Romosozumab Overall
Number analyzed (Participants) | 104 | 214
percent change | 1.87 (0.441) | 4.66 (0.371)

ADVERSE EVENTS:
Time Frame: From Baseline to Safety Follow Up (up to Month 15)
Description: SS - all randomized study participants who received at least 1 dose of IMP. As pre-specified in Protocol and SAP, TEAEs were assessed and reported for 6 months for participants in placebo/romo arm (OL Period) and for a total of 12 months for participants in romo/romo arm (DB Period + OL Period combined) + 3 months of Safety follow-up for both arms (Up to Month 15) during Overall Period. SS for OL period consisted of all randomized study participants who received at least 1 dose of IMP.
Arm/Group | Placebo | Romosozumab | Placebo/Romosozumab | Romosozumab/Romosozumab Overall
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/218 | 0/98 | 1/218
Serious Adverse Events (participants affected / at risk) | 5/109 | 8/218 | 9/98 | 25/218
Other Adverse Events (participants affected / at risk) | 25/109 | 59/218 | 59/98 | 155/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=109) | Romosozumab (N=218) | Placebo/Romosozumab (N=98) | Romosozumab/Romosozumab Overall (N=218)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bone hypertrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=109) | Romosozumab (N=218) | Placebo/Romosozumab (N=98) | Romosozumab/Romosozumab Overall (N=218)
COVID-19 (Infections and infestations) | 12 (12) | 15 (15) | 22 (22) | 49 (50)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 13 (16) | 6 (8) | 30 (37)
Suspected COVID-19 (Infections and infestations) | 4 (4) | 11 (11) | 14 (14) | 43 (43)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 11 (13) | 1 (1) | 22 (25)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 6 (6) | 16 (16)
Nasopharyngitis (Infections and infestations) | 1 (1) | 8 (8) | 2 (3) | 11 (12)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 3 (3) | 3 (3) | 12 (12)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 9 (9) | 4 (4) | 12 (12)
Injection site reaction (General disorders) | 1 (1) | 19 (27) | 6 (9) | 20 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (9) | 1 (1) | 16 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 12 (12) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT05067335/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT05067335/SAP_001.pdf